CLINICAL TRIAL: NCT01109862
Title: Prospective Randomized Comparison of Bipolar Hemiarthroplasty and Total Hip Arthroplasty With Large Femoral Heads for the Treatment of Displaced Intracapsular Femoral Neck Fractures in the Elderly
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Dror Lakstein, MD, Orthopaedic dept, E.Wolfson medical center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0019-10-WOMC
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2010-04

CONDITIONS: Femoral Neck Fractures
Keywords: Femoral neck fractures; Hip fractures; Elderly; Total hip arthroplasty; Bipolar hemiarthroplasty
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures | interventions — Arthroplasty, Replacement, Hip; Hemiarthroplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- THA (Experimental): Total hip arthroplasty
  Interventions: Procedure: Total hip arthroplasty
- HAP (Active Comparator): Bipolar Hemiarthroplasty
  Interventions: Procedure: Hemiarthroplasty

INTERVENTIONS:
Procedure: Total hip arthroplasty — All cemented THA
  Arms: THA
Procedure: Hemiarthroplasty — Cemented bipolar HAP
  Arms: HAP

SUMMARY:
The purpose of this study is to compare hemiarthroplasty (HAP) with total hip arthroplasty (THA), performed by trained arthroplasty surgeons with the use of large femoral heads for the treatment of displaced femoral neck fractures in mobile independent elderly patients, to determine the impact of these surgical options on the short term functional outcomes and complication rates, namely dislocation and the need for further surgery.

This is a single-blinded prospective randomized clinical trial comparing functional outcome and complication rates of 40 patients treated with all cemented THA to a control group of 40 patients treated with cemented bipolar HAP, in a 2 years followup.

The primary endpoint is the Oxford hip score (OHS) at last followup as a measure of functional outcome. Secondary endpoints include the SF-36 score, walking distance and rates of postoperative dislocation, component loosening, need for revision and postoperative mortality.

ELIGIBILITY:
Inclusion Criteria:

* 1. Acute femoral neck fracture.
* 2. Age between 70 and 90 years old.
* 3. Independent community ambulator (more than 0.5km, without the aid of another person. The use of a cane is permitted) prior to fracture.
* 4. Abbreviated mental test score > 6 .

Exclusion Criteria:

* 1. Pathological fracture (excluding osteoporosis).
* 2. Rheumatoid arthritis.
* 3. Symptomatic arthrosis of the involved hip.
* 4. Neurological disorder that may significantly influence walking ability and/or tendency to dislocate.
* 5. Chronic corticosteroid use.
* 6. Concomitant other fracture.
* 7. Very high surgical risk.

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Oxford hip score (OHS) | last followup - 2 years

SECONDARY OUTCOMES:
SF-36 score, walking distance | 2 years followup
dislocation rate, mortality rate | within follow up - 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dror Lakstein, MD, Principal Investigator — E. Wolfson medical center
Locations (1):
- Orthopaedic dept., E. Wolfson Medical center, Holon, Israel

REFERENCES:
- See also: Institutional web site — http://www.wolfson.org.il